CLINICAL TRIAL: NCT06716710
Title: The Effect of the Clinical Activity Applied to High-Risk Pregnant Women on Pregnancy Stress and Fear of Childbirth
Brief Title: Intervention for Fear of Childbirth in High-Risk Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Sena Dilek Aksoy, Principal Investigator, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: sdilek13
Record Dates: First submitted 2024-11-29; First posted 2024-12-04 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Threatened Premature Birth; Premature Membrane Rupture; Gestational Hypertension; Intrauterine Growth Retardation (IUGR); Placenta Previa; Hyperemesis Gravidarum - Severe; Multiple Pregnancy
Keywords: Art Therapy; Fear; High-Risk Pregnancy; Stress
MeSH Terms: conditions — Fetal Membranes, Premature Rupture; Hypertension, Pregnancy-Induced; Fetal Growth Retardation; Placenta Previa | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Art therapy group (Experimental): In addition to the medical treatments that the pregnant women in the study group will receive in the clinic for 4 weeks, they will be given 2 mandala painting sessions, 3 days a week, under the supervision of the researcher.
  Interventions: Behavioral: Art therapy group
- Control group (Other): Nothing other than routine procedures will be done to the control group.
  Interventions: Other: Control group

INTERVENTIONS:
Behavioral: Art therapy group — In addition to the medical treatments that the pregnant women in the study group will receive in the clinic for 4 weeks, a mandala coloring session will be held 3 days a week, 2 times a week under the supervision of the researcher. In order to ensure standardization in the pregnant women included in the study group, each pregnant woman will be given the same mandala work box (36 colored coloring pencils, file, eraser, pencil sharpener and the same mandala prints for all pregnant women). The selection of mandala patterns will be determined by the researchers. In the second week of the training, the researcher will evaluate the STAI TX1 and STAI TX 2, Pregnancy Stress Scale, and FOBS fear of birth scale. At the end of the four-week activity, the researcher will evaluate again.
  Arms: Art therapy group
Other: Control group — In addition to the medical treatments that the pregnant women in the control group will receive in the clinic for 4 weeks, no other application will be made. After two weeks, the researcher will evaluate them using the STAI TX1 and STAI TX 2, Pregnancy Stress Scale, and FOBS fear of childbirth scale. At the end of the fourth week, the researcher will evaluate them again.
  Arms: Control group

SUMMARY:
The aim of the study is to examine the effects of mandala activity applied to pregnant women hospitalized due to high-risk pregnancies on pregnancy stress and fear of childbirth. The study was designed as an experimental study. The sample size of the study was calculated based on the study conducted by Rondung et al. in 2018 to evaluate the effects of internet-based cognitive behavioral therapy on fear of childbirth. The sample size of the study was calculated using G*Power 3.1. 9.2 and the mean and standard deviation values of the effect of cognitive behavioral therapy on fear of childbirth variable in the relevant article were taken into account to calculate the effect size. The blended effect size was calculated as 0.28 using the mean and standard deviation of the relevant article. The minimum number of individuals to be included in the sample of this study was calculated with G*Power 3.1. 9.2 using effect size: 0.28, α= 0.05, power: 0.95 (group1= 75, group2-75) and the sample size was determined to be at least 75 participants in each group. To collect data in the study, Individual Informed Consent Form, Introductory Information Form, STAI FORM TX - 1, STAI FORM TX - 2, Pregnancy Stress Assessment Scale, Fear of Birth Scale will be used.

DETAILED DESCRIPTION:
Aim: The aim of the study is to examine the effect of mandala activity applied to pregnant women hospitalized in the clinic due to high-risk pregnancies on pregnancy stress and fear of birth.

Hypothesis 1 H.0: There is no difference in pregnancy stress scores between high-risk pregnant women who participated in the mandala study applied in addition to medical treatment in the hospital and high-risk pregnant women who did not.

H.1: There is a difference in pregnancy stress scores between high-risk pregnant women who participated in the mandala study applied in addition to medical treatment in the hospital and high-risk pregnant women who did not.

Hypothesis 2 H.0: There is no difference in state scores between high-risk pregnant women who participated in the mandala study applied in addition to medical treatment in the hospital and high-risk pregnant women who did not.

H.1: There is a difference in state scores between high-risk pregnant women who participated in the mandala study applied in addition to medical treatment in the hospital and high-risk pregnant women who did not.

Hypothesis 3 H.0: There is no difference in trait anxiety scores between high-risk pregnant women who participated in the mandala study applied in addition to medical treatment in the hospital and high-risk pregnant women who did not.

H.1.: There is a difference in the trait anxiety scores of high-risk pregnant women who participated in the mandala study applied in addition to medical treatment in the hospital and high-risk pregnant women who did not participate.

Hypothesis 4 H.0.: There is no difference in the childbirth anxiety scores of high-risk pregnant women who participated in the mandala study applied in addition to medical treatment in the hospital and high-risk pregnant women who did not participate.

H.1.: There is a difference in the childbirth anxiety scores of high-risk pregnant women who participated in the mandala study applied in addition to medical treatment in the hospital and high-risk pregnant women who did not participate.

Hypothesis 5. H.0.: There is no difference in the childbirth fear scores of high-risk pregnant women who participated in the mandala study applied in addition to medical treatment in the hospital and high-risk pregnant women who did not participate.

H.1.: There is a difference in the childbirth fear scores of high-risk pregnant women who participated in the mandala study applied in addition to medical treatment in the hospital and high-risk pregnant women who did not participate.

Implementation of the Study The study will be explained to the pregnant women included in the study sample, and informed consent forms and permissions will be obtained from those who voluntarily agree to participate. In the study, an introductory information form, STAI TX1 and STAI TX 2, Pregnancy Stress Scale, and FOBS fear of childbirth scale will be used for pregnant women who are admitted to a public hospital gynecology department in Kocaeli and who meet the research criteria. During the interview, mobile phone numbers will be obtained from the pregnant women for communication purposes, and e-mail addresses will be obtained for participation via online platforms (Zoom, Google Meet, etc.) in order to implement the activities in case they are discharged. The forms required for the follow-up of the pregnant women included in the study and control groups will be presented to the pregnant women in printed form. In addition to the medical treatments they will receive in the clinic for 4 weeks, the pregnant women included in the study group will be given 2 mandala painting activities 3 days a week under the supervision of the researcher. In order to ensure standardization in the pregnant women included in the study group, the same mandala work box (36 colored pencils, file, eraser, pencil sharpener and the same mandala prints for all pregnant women) will be given to each pregnant woman. The selection of mandala patterns will be determined by the researchers. In the second week of the training, the researcher will evaluate using STAI TX1 and STAI TX 2, Pregnancy Stress Scale, FOBS fear of childbirth scale. At the end of the four-week activity, the researcher will repeat STAI FORMTX-1, STAI FORMTX-2, Pregnancy Stress Scale and FOBS fear of childbirth scale to determine the level of pregnancy stress and fear of childbirth in the study and control groups, and the final status of pregnancy stress and fear of childbirth will be evaluated. In the event that the participants are discharged from the clinic, the researcher will implement the activities and evaluate the forms through Online Platforms.

Statistical analysis will be used using IBM SPSS Statistic 29.0 (IBM Corp., Armonk, NY, USA). Compliance with normal distribution will be assessed with Shapiro-Wilk. Descriptive statistical methods will be used in the analysis of sociodemographic data. Categorical data with normal distribution will be assessed with parametric tests (chi square, T test etc.), and those that are not will be assessed with nonparametric tests (Mann-Whitney U Test, Kruskal Wallis etc.). One-Way Analysis of Variance in Repeated Measures will be used in the evaluation of repeated measurements. The significance level will be accepted as p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Those who want to participate in the study voluntarily
* Those who can speak and understand Turkish
* Those who are over 18 years of age
* Primiparous pregnant women
* Pregnant women diagnosed with risky pregnancies (threatened preterm labor, premature rupture of membranes, gestational hypertension, intrauterine growth retardation, placenta previa, hyperemesis gravidarum)
* Pregnant women in the second and third trimesters of pregnancy (13-40 weeks)
* Those who do not have hearing, comprehension and vision problems so that they can follow the group study will be included in the study.

Exclusion Criteria:

* Pregnant women who are absent from the mandala activity planned 3 times a week for 4 weeks for more than a week
* Those who do less than 18 mandala activities during 4 weeks
* Those who fill out the survey forms incompletely
* Pregnant women who decide to give birth during the survey period will be excluded from the study.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 149 (Actual)
Dates: Start 2024-09-16 (Actual); Primary Completion 2025-10-16 (Actual); Study Completion 2025-12-16 (Actual)

PRIMARY OUTCOMES:
State-Trait Anxiety Inventory (STAI FORM TX) | It will be used at the end of the 2nd week and the end of the 4th week of the study.
  It will be used to measure state and trait anxiety.
Pregnancy Stress Scale | It will be used at the end of the 2nd week and the end of the 4th week of the study.
  It will be used to measure the stress of the pregnant woman
Fear of Birth Scale | It will be used at the end of the 2nd week and the end of the 4th week of the study.
  It will be used to measure the fear of childbirth.

CONTACTS AND LOCATIONS:
Overall Officials: Sena Dilek Aksoy, Ph.D., Principal Investigator — Kocaeli University; Sena Ozen, Study Chair — Kocaeli City Hospital
Locations (1):
- Kocaeli University, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rondung E, Ternstrom E, Hildingsson I, Haines HM, Sundin O, Ekdahl J, Karlstrom A, Larsson B, Segeblad B, Baylis R, Rubertsson C. Comparing Internet-Based Cognitive Behavioral Therapy With Standard Care for Women With Fear of Birth: Randomized Controlled Trial. JMIR Ment Health. 2018 Aug 10;5(3):e10420. doi: 10.2196/10420. PMID 30097422